CLINICAL TRIAL: NCT05775900
Title: Efficacy and Safety of Triweekly Cetuximab in Combination With Capecitabine as First-line Maintenance Treatment for KRAS/BRAF Wild-type Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-29
Record Dates: First submitted 2023-02-25; First posted 2023-03-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: First-line Maintenance Therapy; Triweekly Cetuximab; KRAS/BRAF Wild-type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab in Combination With Capecitabine (Experimental): Patients were given cetuximab (a '3+3' design was adopted in the experimental arm, with four dose levels of 400mg/m2, 500mg/m2, 600mg/m2 and 700mg/m2 for dose exploration) every 3 weeks (Q3W).
  Capecitabine, 1000mg/m2, twice a day (BID, once in the morning and once in the evening), 14 days of continuous oral administration followed by 7 days of rest.
  The two-drug combination therapy was continued every 3 weeks in a cycle until patients developed disease progression or met other criteria for termination of study treatment specified in the protocol.
  Interventions: Drug: Cetuximab; Drug: Capecitabine

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be given triweekly at a dose from 400mg/m2 to 700mg/m2.
  Other Names: Erbitux
Drug: Capecitabine — Capecitabine will be given 2 weeks on/1 week off (1000mg/m2 BID po.)
  Other Names: Capecitabine Tablets

SUMMARY:
To explore the safety, efficacy and pharmacokinetic (PK) characteristics of triweekly cetuximab in combination with capecitabine as first-line maintenance treatment for KRAS/BRAF wild-type metastatic colorectal cancer: a single-arm, a single-center, Phase 1b trial. Meanwhile, Exploring the maximum tolerant dose or recommended II research dose of triweekly cetuximab combined with a fixed dose of capecitabine using '3+3' dose climbing Phase I experiment.

ELIGIBILITY:
Inclusion Criteria:

* Provide a written informed consent form (ICF) before any research procedure is carried out.
* Patients must be ≥18 years old and have an expected life span of at least 12 weeks when signing the ICF.
* Patients have histologically or cytologically confirmed RAS and BRAF wild-type metastatic colorectal adenocarcinoma (mCRC), excluding appendiceal and anal cancers.
* After being diagnosed with mCRC, patients have only received cetuximab combined with chemotherapy (FOLFOX or FOLFIRI) as first-line induction therapy. Imaging progression during adjuvant therapy or within 6 months after completion of adjuvant therapy is considered as first-line treatment.
* Patients have completed 8 cycles of cetuximab combined with chemotherapy induction therapy and the disease is controlled (including CR/PR and SD).
* There is at least one measurable metastatic lesion, defined as per RECIST version 1.1. Patients who have achieved CR without measurable lesions after induction therapy, and those who have achieved no evidence of disease (NED) through R0 resection, interventional ablation, or other local destructive therapies can be included in this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Within 7 days before treatment, the following laboratory test values are obtained and appropriate organ function is present:

Hemoglobin ≥ 90g/L, neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 75 × 10^9/L; Serum total bilirubin ≤ 1.5 × upper limit of normal (UNL); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × UNL; if there are liver metastases, AST or ALT ≤ 5 × UNL; Serum creatinine ≤ 1.5 × UNL.

* Patients are not allowed to participate in other clinical trials during the study period.
* Patients are willing and able to comply with the study protocol and visit plan.

Exclusion Criteria:

* Excluding adjuvant therapy that ended more than 9 months ago (including oxaliplatin-containing therapy) or more than 6 months ago (excluding oxaliplatin-containing therapy), any chemotherapy for metastatic colorectal cancer (mCRC) other than induction therapy consisting of cetuximab in combination with FOLFOX or FOLFIRI.
* Concurrent active malignancy, excluding malignancies with disease-free survival of 5 years or more or in situ carcinoma considered cured after adequate treatment.
* Known brain metastases or leptomeningeal metastases. Patients with neurological symptoms should undergo brain CT/MRI to exclude metastases.
* Any unresolved toxicities greater than or equal to Grade 2 per the Common Terminology Criteria for Adverse Events (CTCAE) caused by previous treatment, excluding alopecia, skin pigmentation, and anemia. Patients with unresolved neurotoxicity greater than or equal to CTCAE Grade 3 caused by platinum-based drugs should be excluded.
* Ascites, pleural effusion, or pericardial effusion requiring drainage within the past 4 weeks.
* Patients with bowel obstruction, gastrointestinal bleeding, pulmonary fibrosis or interstitial pneumonia, renal failure, liver failure, or cerebrovascular disease.
* Uncontrolled diabetes, defined as HbA1c >7.5% after the use of antidiabetic drugs, or uncontrolled hypertension, defined as systolic/diastolic blood pressure >140/90mmHg after the use of antihypertensive drugs.
* Myocardial infarction within the past 12 months, severe/unstable angina pectoris, or New York Heart Association (NYHA) Class III or IV congestive heart failure symptoms.
* A history of allergy to any study drugs (such as cetuximab or capecitabine).
* Known infection with human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS) related diseases, hepatitis B or C.
* Autoimmune diseases or a history of organ transplantation requiring immunosuppressive therapy.
* Mental illness that may increase the risk associated with participation in the study or interfere with the interpretation of study results.
* Received any of the following treatments within a specified time period prior to receiving the study drug:

Major surgery within 4 weeks (excluding diagnostic biopsy, surgical incision should be completely healed before administering the study drug).

Radiotherapy within 4 weeks. Other anti-tumor treatments or participation in other clinical trials within 4 weeks, except for induction therapy as specified in the protocol.

* Pregnant (confirmed by serum human chorionic gonadotropin [hCG] test) or lactating women, or women of childbearing potential who plan to become pregnant during the treatment period and within 2 months after the end of cetuximab treatment, or within 6 months after the end of capecitabine treatment. Women of childbearing potential or sexually active men who are unwilling to use contraception during the study period and for at least 2 months after the end of cetuximab treatment, or 6 months after the end of capecitabine treatment. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Presence of any other serious illness that, in the investigator's opinion, would preclude the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Safety variables (Incidence of Adverse Events [Safety and Tolerability]) | 2 year
  Safety variables will be summarized using descriptive statistics based on adverse events collection
Pharmacokinetic (PK) characteristics 1 | 2 year
  Evaluation Peak Concentration (Cmax) of cetuximab before and after Treatment.
Pharmacokinetic (PK) characteristics 2 | 2 year
  Evaluation Area Under the Curve (AUC0-t, AUC0-∞) of cetuximab before and after Treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 year
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first. When a patient was alive and without progression, PFS was censored at the date of the last disease assessment.
Overall Survival (OS) | 2 year
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Objective response rate (ORR) | 2 year
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR).
Disease Control Rate (DCR) | 2 year
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Quality of Life (QOL) | 2 year
  Evaluation of alterations in patients' quality of life throughout treatment by using the EORTC QLQ-CR29 and EORTC QLQ-CR30 quality of life questionnaire. Evaluation of the scores was based on the Karnofsky Performance Scale (KPS). The reliability and validity of the questionnaires were assessed by Cronbach's α coefficient, the Spearman correlation test and Wilcoxon rank sum test.

OTHER OUTCOMES:
Treatment-emergent genetic mutations | 2 year
  Assessment of the correlation between mutation status of relevant genes and treatment response through ctDNA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China